CLINICAL TRIAL: NCT03212118
Title: Effects of Motivational Interviewing for Long-term Sick Absence: A Randomized Controlled Trial With Mixed Methods
Brief Title: Effects of Motivational Interviewing for Long-term Sick Absence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University of Bergen (Other); University of Oslo (Other); National Center for Occupational Rehabilitation, Rauland (Unknown); Deakin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/2300-C
Record Dates: First submitted 2017-06-12; First posted 2017-07-11 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Sick Leave
Keywords: Sick Leave; Return to work; Motivational interviewing; Absenteeism; Occupational Health
MeSH Terms: interventions — Therapeutics; Motivational Interviewing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment as usual (Other): Treatment as usual "untouched". This is the standard The Norwegian Labour and Welfare Administration (NAV) procedure.
  Interventions: Behavioral: Treatment as usual (TAU-0)
- Two talks (Active Comparator): Two standard talks (not including elements from motivational interviewing)
  Interventions: Behavioral: Structured talks (TAU-2)
- Motivational interviewing (Experimental): Two standard talks with a motivational interviewing content.
  Interventions: Behavioral: motivational interviewing (MI)

INTERVENTIONS:
Behavioral: Treatment as usual (TAU-0) — The standard NAV procedure, which consists of a telephone call within 8 weeks to an employer who have employees on 100% sick leave, in addition to regular NAV conversations "on-demand" (not "fixed intervals") between the NAV caseworkers and the employees.
  Other Names: 'untouched'
  Arms: Treatment as usual
Behavioral: Structured talks (TAU-2) — Two structured talks (not including elements from motivational interviewing)
  Other Names: non-MI
  Arms: Two talks
Behavioral: motivational interviewing (MI) — Two structured talks (must have a valid motivational interviewing content).
  Other Names: MI
  Arms: Motivational interviewing

SUMMARY:
Long-term sickness absence has considerable impact on social functioning, families involved, the employer, and society as a whole. Preventing long-term sickness absence and increase the likelihood of return to work (RTW) are critical concerns for industrialized countries across the world. Motivational factors contributing to RTW and maintenance of work participation are therefore of importance to explore in order to get the person back to work after long-term sick leave. Motivational interviewing (MI) is an empirically validated psychological approach that may be particularly useful in a RTW context. Even though MI has been widely studied and is considered a flexible intervention strategy in different domains, its effectiveness in improving RTW has not yet been studied.

The aim of this study is to evaluate whether MI provided by trained caseworkers at The Norwegian Labour and Welfare Administration (NAV) to sick-listed users with unselected diagnoses facilitates RTW compared with follow-up as usual.

DETAILED DESCRIPTION:
The main study will be preceded by a pilot study (anticipated start medio august 2017). The aim of the pilot is to test the practical aspects of the study. If no changes are made to the study protocol, the intervention or one of the other arms, participants from the pilot will be included in the main study, In case of modifications to the study protocol after the pilot, participants from the pilot study will not be included in the main study. Data for primary and secondary outcomes will not be assessed before the end of the main study.

In addition to the intention to treat and per protocol analyses, subgroup analyses will be performed if sufficient power for age, gender, diagnoses for sick leave, occupational category and length of previous sick leave.

In addition to the effect evaluation, qualitative studies, a feasibility/process evaluation study and a health economic evaluation (cost-effectiveness, cost-utility and cost-benefit) will be performed. The qualitative studies will be based on data from focus group discussions. The main areas for investigation will be:

* The participants' expectations to return to work before and after motivational interviewing.
* Perceived facilitators and obstacles for return to work among participants
* The perceived benefits and challenges in using motivational interview to facilitate a return to work process

Changes made Sept.29 2017: Due to slow recruitment, it was decided to leave out one of the arms from the study (TAU-1: extra phone call to employer). The extra phone call element was also taken out from the other arms where it was included. Another reason for this change was that the TAU-1 intervention arm was not ideally designed to evaluate the extra phone call. It was decided this intervention arm is better evaluated in a separate trial. Currently 12 persons are included and randomized in the trial. Those who are randomized to TAU-1 and have not received an intervention, will be randomized again. The ones randomized to TAU-1 who already have got an intervention will stop participating in the study.

Changes made Aug. 26 2019: Due to problems with implementation of the intervervention the first couple of months, it was decided to start inclusion from Jan 1st 2018 (instead of Aug 2017). The planned number of participants has not changed.

Clarification added April 25 2021. Regarding exclusion criterion unemployment: only sick listed individuals listed with an employer were identified in the sick leave registries and invited to take part in the study. That means individuals who were unemployed, self-employed or for other reasons without an employer were not included.

ELIGIBILITY:
Inclusion Criteria:

* Living in the county Sør-Trøndelag
* On sick leave for 8 weeks
* Current sick leave status of 50-100%

Exclusion Criteria:

* no employment
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 774 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Total number of sickness absence days during the year after enrollment in the study (i.e. after randomization) | 12 months
  Register data from the national health and welfare services

SECONDARY OUTCOMES:
The time until full sustainable return to work (RTW), i.e. for at least 4 weeks without relapse | 12 months
  Register data from the national health and welfare services
Probability of working (i.e. not receiving medical benefits) each month during follow-up, measured as repeated events | 12 months
  Register data from the national health and welfare services
Return to Work Self-Efficacy | 12 months
  Return to Work Self-Efficacy Scale (Lagerveld et al, 2010)
Resilience | 12 months
  Resilience Scale for Adults (Friborg et al, 2003)
Return to work expectations | 12 months
  Expectations about length of sick leave and return to work (3 items)
Workability | 12 months
  Single question. How will you rate your work ability (scale from 0 (no ability) to 10 (my best ability)) (1 item)
Health-related quality of life | 12 months
  EQ- 5D- 5L Questionnaire, Herdman et al, 2011

OTHER OUTCOMES:
Pain | 12 months
  Brief Pain Inventory (BPI), 1 item
Fatigue | 12 months
  Fatigue Severity Scale (FFS), 1 item
Sleep problems | 12 months
  Insomnia Severity Index, 5 items
Anxiety symptoms | 12 months
  Generalized Anxiety Disorder 7-item (GAD-7)
Depression symptoms | 12 months
  Patient Health Questionnaire (PHQ-9)

CONTACTS AND LOCATIONS:
Overall Officials: Egil Andreas Fors, phd prof, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Dept, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No
Individual data will not be available for other researchers due to ethical approval.

REFERENCES:
- [Background] Aasdahl L, Foldal VS, Standal MI, Hagen R, Johnsen R, Solbjor M, Fimland MS, Fossen H, Jensen C, Bagoien G, Halsteinli V, Fors EA. Motivational interviewing in long-term sickness absence: study protocol of a randomized controlled trial followed by qualitative and economic studies. BMC Public Health. 2018 Jun 18;18(1):756. doi: 10.1186/s12889-018-5686-0. PMID 29914463
- [Derived] Foldal VS, Solbjor M, Standal MI, Fors EA, Hagen R, Bagoien G, Johnsen R, Hara KW, Fossen H, Lochting I, Eik H, Grotle M, Aasdahl L. Barriers and Facilitators for Implementing Motivational Interviewing as a Return to Work Intervention in a Norwegian Social Insurance Setting: A Mixed Methods Process Evaluation. J Occup Rehabil. 2021 Dec;31(4):785-795. doi: 10.1007/s10926-021-09964-9. Epub 2021 Mar 24. PMID 33761083
- [Derived] Foldal VS, Standal MI, Aasdahl L, Hagen R, Bagoien G, Fors EA, Johnsen R, Solbjor M. Sick-listed workers' experiences with motivational interviewing in the return to work process: a qualitative interview study. BMC Public Health. 2020 Feb 28;20(1):276. doi: 10.1186/s12889-020-8382-9. PMID 32111199

DOCUMENTS (1):
  • Statistical Analysis Plan (2020-03-30): https://cdn.clinicaltrials.gov/large-docs/18/NCT03212118/SAP_000.pdf